CLINICAL TRIAL: NCT04410848
Title: Symbolic Regression Model To Predict Choledocholithiasis: Prospective Validation
Brief Title: Symbolic Regression Model To Predict Choledocholithiasis
Acronym: (SymChole)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med. Hector Eloy Tamez Perez, Clinical Professor, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: GA19-00003
Record Dates: First submitted 2020-01-20; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Common Bile Duct Calculi
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patient with suspicion of choledocholithiasis: Patient with the suspect of common biliary duct stone for pain type colic in the right upper quadrant abdomen, the elevation of bilirubin, alkaline phosphatase, pancreatitis, dilated common bile duct and cholangitis. According to the criteria to assign the risk of choledocholithiasis. We are going to validate a scale based on intelligence artificial compared to the clinical predictor.
  Interventions: Other: To determine the diagnostic of Choledocholithiasis with symbolic regression model

INTERVENTIONS:
Other: To determine the diagnostic of Choledocholithiasis with symbolic regression model — To determine the diagnostic of Choledocholithiasis with symbolic regression model

SUMMARY:
Choledocholithiasis refers to the presence of gallstones within the common bile duct. It is proposed to look for markers that help in the diagnosis and in differentiating between retained and migrated gallstones. The selection of patients is a very important aspect, due to the economic aspects and possible complications. Taking advantage of the development of technology, the improvement in computer systems, the use of artificial intelligence and a symbolic regression model that works to predict the presence of choledocholithiasis and provide evidence that clarifies the treatment of patients with this pathology, especially in this group where there is a bigger controversy.

DETAILED DESCRIPTION:
Choledocholithiasis refers to the presence of gallstones within the common bile duct. It is proposed to look for markers that help in the diagnosis and in differentiating between retained and migrated gallstones. The selection of patients to perform endoscopic retrograde cholangiopancreatography (ERCP) is a very important aspect, due to the economic aspects and possible complications. By making a proper patient selection for additional studies or procedure, then the costs, complications and days of stay would be reduced. Avoiding the unnecessary use of ERCP would avoid its complications. Taking advantage of the development of technology, the improvement in computer systems, the use of artificial intelligence and a Symbolic Regression Model that works to predict the presence of choledocholithiasis and provide evidence that clarifies the treatment of patients with this pathology, especially in this group where there is a bigger controversy.

Having the historical database of the University Hospital (HU), regarding clinical, laboratory and image variables of patients with suspected choledocholithiasis, using a symbolic regression method, several randomly formed equations are generated. Each equation deducts its coefficient of linear correlation (Pearson's correlation).

For the following study we admitted to the emergency department of adults at the University Hospital all patients with clinical suspicion of choledocholithiasis, who meet the inclusion criterion. The study which is realized is a normal one based on the method of clinical predictors, obtaining laboratory studies, image studies, and patient management will be carried out based on the method of clinical predictors. The calculation is made with the equation obtained, and the patient is monitored until discharge. The calculation obtained from the equation will not be taken into account for the decisions in the management of the patient. The variables studied as white blood cells, total bilirubin values, direct bilirubin, indirect bilirubin, Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST), alkaline phosphatase (AP), gamma-glutamyl transpeptidase (GGT) at admission will be taken from the clinical record. Transabdominal ultrasonography will be performed upon admission by the diagnostic radiology department of the HU and the size of the bile duct in mm, presence of gallbladder gallstones and bile duct stones will be taken from the report. ERCP, magnetic resonance cholangiopancreatography (MRCP) or intraoperative cholangiography will be performed and one will be taken as a confirmation of choledocolithiasis, and its absence would rule it out.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 with clinical suspicion of choledocholithiasis by biliary-type pain, laboratory testing that reveals a cholestatic pattern of liver test abnormalities, biliary pancreatitis or dilated common bile duct

Exclusion Criteria:

* Patient with a history of cholecystectomy
* History of previous ERCP or surgery involving bile duct
* Patient who could not be followed
* Patient with other pathology that causes alteration of liver function test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical suspicion of choledocholithiasis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
To validate prospectively a symbolic regression model to predict choledocholithiasis | 72 horas
  To validate a model to predict choledocholithiasis compared clinical predictors.

CONTACTS AND LOCATIONS:
Overall Officials: José A. González González, MD, Study Director — José Eleuterio González University Hospital
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez, Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No